CLINICAL TRIAL: NCT03421067
Title: Are we Supporting the Apex During Hysterectomy for Pelvic Organ Prolapse: A NSQIP Analysis.
Brief Title: Apical Support During Hysterectomy for Pelvic Organ Prolapse-NSQIP Analysis.
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 17-111
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective descriptive study using the American College of Surgeon's National Surgical Quality Improvement Program® (ACS NSQIP®) data to determine whether gynecologic surgeons are already meeting the recently recommended best practice of supporting the vaginal apex at time of hysterectomy for pelvic organ prolapse (POP).

DETAILED DESCRIPTION:
The prevalence of pelvic organ prolapse (POP) in the United States is estimated to be between 40-50% with an anticipated increase over the next several decades. Approximately 300,000 women undergo surgeries to repair POP in the United States every year. Following pelvic reconstructive surgery, recurrence rates of symptomatic prolapse range between 6-30%.

Our understanding of pelvic anatomy and its support has been significantly improved over recent decades, with many researchers reporting on details and mechanics previously not understood.

In November 2017, the American College of Obstetricians and Gynecologists released a new practice bulletin outlining the current standard of care for the treatment of women with pelvic organ prolapse. In this bulletin, they state that a hysterectomy alone is not adequate treatment for POP, and further that any woman having a hysterectomy for POP should undergo a concurrent apical suspension procedure as a standard of care.

The purpose of this study is to determine the proportion of patients undergoing hysterectomy for the indication of POP having concurrent apical suspension among the population whose cases are reported within the NSQIP database, and who underwent hysterectomy between 2015 and 2017.

ELIGIBILITY:
Inclusion Criteria:

* Underwent hysterectomy for pelvic organ prolapse, between 2015 and 2017

Exclusion Criteria:

* Age < 18 years old
* Pelvic Organ Prolapse was not recorded in their postoperative diagnoses

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent hysterectomy for pelvic organ prolapse between 2015 and 2017, and whose cases are reported within ACS NSQIP®.
Sampling Method: Non-Probability Sample
Enrollment: 3458 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
proportion of patients having concurrent apical suspension performed | procedure (at time of hysterectomy for pelvic organ prolapse)
  proportion of patients who had concurrent apical support procedures performed

CONTACTS AND LOCATIONS:
Overall Officials: Catrina Crisp, MD, MSc, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates
Locations (1):
- TriHealth - Cincinnati Urogynecology Associates, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No